CLINICAL TRIAL: NCT03256383
Title: Plan for Testing Fingerstick Bloods on Magellan Systems
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Magellan Diagnostics (Industry)
Responsible Party: Sponsor
Other Study IDs: 276
Record Dates: First submitted 2017-08-18; First posted 2017-08-22 (Actual); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Lead Poisoning
MeSH Terms: conditions — Lead Poisoning

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Adult: Patients aged 18+ years
  Interventions: Device: Lead testing
- Children 7 - 17: Patients aged 7 - 17 years
  Interventions: Device: Lead testing
- Children <7: Patients aged under 7 years
  Interventions: Device: Lead testing

INTERVENTIONS:
Device: Lead testing — Fingerstick

SUMMARY:
This study is to supplement our internal data that demonstrates the continued performance of capillary blood samples on Magellan's lead testing systems: LeadCare II, LeadCare Ultra (which have been cleared previously by FDA), and PediaStat, which is an upgraded LeadCare II instrument in development.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects who consent to a capillary blood collection

Exclusion Criteria:

* Patients are not currently taking chelating agents, e.g., penicillamine, succimer

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: adults and children up to 18 years of age who are at risk of lead exposure, pregnant women who are at risk of lead exposure,
Sampling Method: Probability Sample
Enrollment: 190 (Estimated)
Dates: Start 2017-07-31 (Actual); Primary Completion 2017-08-31 (Estimated); Study Completion 2017-08-31 (Estimated)

PRIMARY OUTCOMES:
Lead poisoning | 1 day
  >10ug/dL lead in whole blood is considered lead poisoning These measurements will be taken to compare the fingerstick data collected in the field with data received through reference method

CONTACTS AND LOCATIONS:
Overall Officials: Peter Rappo, MD, Principal Investigator
Locations (3):
- United States (3):
  - Pediatric Associates, Inc., Brockton, Massachusetts
  - Pediatrics Associates, Inc, Hanson, Massachusetts
  - Pediatrics Associates, Inc, West Bridgewater, Massachusetts

DOCUMENTS (2):
  • Informed Consent Form (2017-07-21): https://cdn.clinicaltrials.gov/large-docs/83/NCT03256383/ICF_000.pdf
  • Study Protocol (2017-07-12): https://cdn.clinicaltrials.gov/large-docs/83/NCT03256383/Prot_001.pdf